CLINICAL TRIAL: NCT07181369
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Tolerability, Pharmacokinetic, Pharmacodynamic, and Preliminary Efficacy Trial of GTX-B001 in Healthy Volunteers (Part A) and Patients With Chronic Inducible Urticaria (Part B)
Brief Title: A Phase 1 Study of GTX-B001 in Healthy Subjects and Patients With Chronic Inducible Urticaria
Acronym: CHILL-MC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Granular Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GRN-GTXB001-001; 2025-522126-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects; Cold Urticaria; Symptomatic Dermographism; Chronic Inducible Urticaria
Keywords: Urticaria; Skin diseases; Mast cells; Bispecific antibody; GTX-B001; Infusion; Single Ascending Dose; Healthy subjects; Safety; Pharmacokinetics; Pharmacodynamics; Cold urticaria; Intravenous; symptomatic dermographism
MeSH Terms: conditions — Cold Urticaria; Familial dermographism; Chronic Inducible Urticaria; Urticaria; Skin Diseases | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A (HV) - GTX-B001 (Experimental): Healthy participants will receive a single dose of GTX-B001
  Interventions: Drug: GTX-B001
- Part A (HV) - Normal Saline (Placebo Comparator): Healthy participants assigned to receive placebo will receive a single dose of normal saline
  Interventions: Drug: Normal Saline
- Part B (ColdU/SD) - GTX-B001 (Experimental): Patients with cold urticaria or symptomatic dermographism will receive a single dose of GTX-B001
  Interventions: Drug: GTX-B001
- Part B (ColdU/SD) - Normal Saline (Placebo Comparator): Patients with cold urticaria or symptomatic dermographism assigned to receive placebo will receive a single dose of normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: GTX-B001 — Single infusion of one of up to five dosages of GTX-B001
  Other Names: ALY-301
  Arms: Part A (HV) - GTX-B001; Part B (ColdU/SD) - GTX-B001
Drug: Normal Saline — Single infusion of normal saline
  Arms: Part A (HV) - Normal Saline; Part B (ColdU/SD) - Normal Saline

SUMMARY:
This is a first-in-human study aimed at determining the safety of a single dose of GTX-B001 in healthy participants and in people with chronic inducible urticaria.

DETAILED DESCRIPTION:
GTX-B001 is a humanized bispecific antibody than binds with one arm to a protein called c-Kit and with the second arm to a protein called CD203c, both expressed on mast cells.

This study is a randomized, double-bind, placebo-controlled phase 1 study evaluating the safety, pharmacokinetics and pharmacodynamics of a single dose of GTX-B001 in healthy participants (Part A) and in patients with chronic inducible urticaria (cold urticaria and symptomatic dermographism) who remain symptomatic despite treatment with antihistamines (Part B). In part B, the preliminary efficacy of GTX-B001 on the signs and symptoms of chronic inducible urticaria will also be evaluated.

48 healthy participants are estimated to be enrolled in part A in five ascending cohorts, while 24 patients with chronic inducible urticaria are estimated to be enrolled in Part B in two ascending cohorts.

Potential participants will be screened for up to 4 weeks prior to enrollment. GTX-B001 will be administered intravenously on Day 1 to randomized participants who will be followed for 12 weeks post-treatment.

Participants will be required to attend a total of 9 visits including the screening visit.

ELIGIBILITY:
Key inclusion Criteria (Part A):

* The subject is between 18 and 55 years of age (both inclusive) at the date of screening.
* The subject is in good general health based on the medical history, physical examination and the results of vital signs, electrocardiogram and clinical laboratory, as judged by the investigator.

Key inclusion Criteria (Part B):

* The subject is between 18 and 75 years of age (both inclusive) at the date of screening
* A history of signs and/or symptoms of ColdU or SD experienced ≥ 3 months prior to screening.
* For ColdU patients, a positive provocation test during screening and baseline, using the TempTest® device.
* For SD patients, a positive provocation test with at least 3 pins during screening and baseline, using the FricTest® device.
* Inadequate control of ColdU or SD by second generation H1-antihistamine (sgAH) as defined as the presence of itch and hives following a trigger (e.g. cold or scratching, respectively) within the last 6 weeks prior to screening in spite of use of a sgAH.
* A Urticaria Control Test (UCT) score of < 12 at screening.

Key exclusion Criteria (Parts A & B):

* Presence of any clinically significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, or endocrine disease or disorder that would interfere with the patient's safety or the interpretation of trial results in the judgment of the investigator.
* Treatment with an investigational drug or intervention for any condition within three months of screening, or concurrent participation in another clinical trial in which an investigational drug is administered.
* Treatment with immunomodulating therapy (e.g., intravenous or intramuscular immunoglobulins, systemic corticosteroids, cyclosporine, methotrexate, dapsone, cyclophosphamide, tacrolimus, mycophenolate mofetil, hydroxychloroquine, infliximab, adalimumab, etanercept, etc.) within 4 weeks (or 5 half-lives, whichever is longer) prior to screening.
* Use of any monoclonal antibody or therapeutic protein within 4 weeks (or 5 half-lives, whichever is longer) prior to screening.
* History of anaphylaxis, autoimmune disorders requiring more than topical medication, or asthma requiring regular use of inhaled medication within the past 5 years, unless, in the opinion of the Investigator, the condition is not considered clinically significant and is unlikely to affect subject safety or study outcomes.

Additionally for Part B:

* Disease with symptoms of urticaria or angioedema other than Chronic Urticaria (CU), for example urticaria vasculitis, erythema multiforme, mastocytosis, or drug-induced urticaria. Patients with concomitant Chronic Spontaneous Urticaria (CSU) or other forms of Chronic Inducible Urticaria (CIndU) are eligible provided that symptoms at screening are consistent with ColdU or SD and that ColdU or SD is the dominant form of CU.
* Any other skin disease associated with chronic itching that might influence in the investigators' opinion of the study evaluations and results, e.g., atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, or psoriasis.
* Receipt of any biologic therapy for urticaria control (e.g. omalizumab, dupilumab, ligelizumab, etc.) within three months of screening (whether on-label or off-label).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the incidence and severity of adverse events (Parts A and B) | Day 1 to Day 85
  Safety and tolerability of a single intravenous infusion of GTX-B001 as assessed by the percentage of subjects at each dose level with Grade 2 or higher adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
GTX-B001 pharmacokinetics (Parts A and B) | Day 1 to Day 85
  Serum concentrations of GTX-B001 at specified visits

OTHER OUTCOMES:
GTX-B001 pharmacodynamics (Parts A and B) | Day 1 to Day 85
  Change from baseline in blood biomarkers such as serum tryptase
GTX-B001 pharmacodynamics in skin (Part B) | Day 1 to Day 29
  Change from baseline in mast cell density and mast cell activation markers upon cold or friction provocation, assessed from skin punch biopsy at baseline and three times post-treatment.
Evaluation of immunogenicity (Parts A and B) | Day 1 to Day 85
  Incidence of anti-drug antibodies
Disease control (Part B ColdU) - Critical Temperature Threshold (CTT) | Day 1 to Day 85
  Change from baseline and percentage of responders in Critical Temperature Threshold (CTT) over time as determined by provocation testing using the TempTest®. The CTT determines the highest temperature that induces symptoms.
Disease control (Part B SD) - Critical Friction Threshold (CFT) | Day 1 to Day 85
  Change from baseline and percentage of responders in Critical Friction Threshold (CFT) over time as determined by provocation testing using the FricTest®. The CFT determines the shortest pin length (or lowest pressure) that induces symptoms.
Disease control (Part B) - Urticaria Control Test (UCT) | Day 1 to Day 85
  Change from baseline and percentage of responders for the Urticaria Control Test (UCT). Total score ranges from 0 to 16. A score of 12 or higher indicates well-controlled chronic urticaria, while a score below 12 suggests poorly controlled disease.
Disease control (Part B ColdU) - Cold Urticaria Activity Score (Cold UAS) | Day 1 to Day 85
  Change from baseline in Cold Urticaria Activity Score (Cold UAS). The total score ranges from 0 to 6, the higher the score the higher the disease activity.
Disease control (Part B SD) - Symptomatic Dermographism Activity Score (SDAS) | Day 1 to Day 85
  Change from baseline in Symptomatic Dermographism Activity Score (SDAS)
Disease control (Part B ColdU) - Cold Urticaria Quality of Life Questionnaire (ColdU-QoL) | Day 1 to Day 85
  Change from baseline in Cold Urticaria Quality of Life Questionnaire (ColdU-QoL). The total score ranges from 0 to 100, the higher the score the higher the impairment.
Disease control (Part B SD) - Symptomatic Dermographism Quality of Life Questionnaire (SD-QoL) | Day 1 to Day 85
  Change from baseline in Symptomatic Dermographism Quality of Life Questionnaire (SD-QoL). The total score ranges from 0 to 100, the higher the score the higher the impairment.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Charité Research Organization gmbh, Berlin
  - Fraunhofer Institute For Translational Medicine And Pharmacology, Berlin

IPD SHARING:
Plan to Share IPD: No